CLINICAL TRIAL: NCT01158430
Title: Treatment of Patients With Health Anxiety. A Randomized Controlled Trial of Acceptance and Commitment Therapy (ACT) Group Treatment Compared to a Waiting List
Brief Title: Acceptance and Commitment Group Therapy (ACT) for Patients With Health Anxiety
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001001
Record Dates: First submitted 2010-02-16; First posted 2010-07-08 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Hypochondriasis; Somatization Disorder
Keywords: Hypochondriasis; Acceptance and Commitment Therapy; ACT
MeSH Terms: conditions — Hypochondriasis; Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT group therapy (Experimental): Third generation cognitive behavioral therapy
  Group therapy (ACT) in groups of 9 patients in 9 weekly 3.5-hours sessions & 1 booster session 1 month after 9th session, a total of 35.5 hours
  Interventions: Behavioral: ACT group therapy
- Control (No Intervention): Control group assigned to wait list (treatment as usual). After 9 months they are offered ACT group therapy, but not as part of the research project.

INTERVENTIONS:
Behavioral: ACT group therapy — Group therapy (ACT) in groups of 9 patients in 9 weekly 3.5-hours sessions & 1 booster session 1 month after 9th session, a total of 35.5 hours
  Other Names: Third generation cognitive behavioral therapy
  Arms: ACT group therapy

SUMMARY:
The purpose of this study is to determine the effect of Acceptance and Commitment Therapy (ACT) in groups on functional level, emotional problems, and use of health care in patients with severe health anxiety in a randomized, controlled design.

DETAILED DESCRIPTION:
Health anxiety disorder or Hypochondriasis is a prevalent somatoform disorder, but a rarely used diagnosis in clinical practice despite studies having reported prevalence between 0.8-9.5% in primary care (Fink et al, 2004). As a consequence, the disorder is rarely treated.

The lack of valid, reliable, and generally accepted diagnostic criteria has been a major obstacle in clinical practice and Hypochondriasis studies, which causes problems particularly in distinguishing Hypochondriasis patients from other patients presenting with medically unexplained symptoms or functional symptoms.

In 2004, the investigators introduced a radically revised definition of Hypochondriasis. Hypochondriasis is viewed as a stigmatizing label, and the designation health anxiety has been suggested as replacement. This new diagnosis is empirically established. The essential feature of health anxiety is that the patients present with cognitive symptoms such as unfounded worrying about their health. In contrast to other somatoform disorders, the patients are not necessarily plagued by physical symptoms.

The new diagnostic criteria include the symptom 'obsessive rumination about illness' plus at least one of the symptoms 'worry or preoccupation with fears of harboring an illness or with bodily functions', 'suggestibility or autosuggestibility', 'an unrealistic fear of being infected or contaminated', 'an excessive fascination with medical information', or 'fear of taking prescribed medication'.

In the current study, health anxiety is diagnosed by use of newly introduced empirically established positive criteria for Health anxiety (Fink et al, 2004).

Most patients with health anxiety disorder receive the majority of their care in primary care settings. They are often unhappy with the services they receive, and primary care providers often feel unprepared to address symptoms that primarily appear functional.

During the past 5 years, the investigators have treated patients suffering from severe functional disorder (i.e. Bodily distress syndrome or Somatization disorder) in randomized controlled trials (RCTs) - at the Research Clinic. The investigators reject many patients suffering from health anxiety, who have no other treatment opportunities, and there is an impending need for treatment opportunities. The investigators research group has done research in epidemiology, psychopathology and diagnostics of Health anxiety, and the investigators are part of international networks regarding the revision of the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders V (DSM-V) and the International Classification of Diseases 11 (ICD-11).

RCTs have shown that Cognitive Behavioral Therapy (CBT) has effect on health anxiety (Barsky & Ahern, 2004; Greeven et al., 2007), and one of the trials also showed effect of anti-depressant medication (Greeven et al., 2007).

In general, the treatment of health anxiety is sparsely investigated both as to psychotherapy and medical treatment.

The investigators wish to examine the effect of Acceptance and Commitment Therapy (ACT) in groups on functional level, emotional problems, and use of health care in patients with severe health anxiety in a randomized, controlled design.

Health anxiety disorder is a burden for the sufferers and costly for society due to lost working years because of early onset of the disorder and high health care costs. The development of evidence-based treatment offering these patients the same professional treatment as patients with other disorders may lead to better quality of life for the patients and reduction in health care costs.

ELIGIBILITY:
Inclusion Criteria:

1. Whiteley-7 score on 21,4 or more (scale 0-100 score points).
2. Severe health anxiety (diagnosed by SCAN interview).
3. Age 20-60 years
4. Patients of Scandinavian origin who understand, read, write and speak Danish.
5. No lifetime-diagnosis of psychoses, bipolar affective disorder or depression with psychotic symptoms (ICD-10: F20-29, F30-31, F32.3, F33.3)
6. In case of a co morbid functional or other psychiatric disorder health anxiety must be the dominating problem.

Exclusion criteria:

1. Another severe psychiatric disorder or if the patient is suicidal.
2. Abuse of narcotics or alcohol and (non-prescribed) medicine.
3. Pregnancy.
4. No informed consent.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Health anxiety measured by the Whiteley-7 index | 9 months (2nd follow-up)

SECONDARY OUTCOMES:
Social level of functioning measured with Short Form health status questionnaire from the medical outcome status (SF-36) | 9 months (2nd follow-up)
Social level of functioning, emotional disorders measured with relevant sub-scales from Symptom Check List, 90 items (SCL 90) | 9 months (2nd follow-up)
Social level of functioning measured with an alcohol dependency questionnaire (CAGE) | 9 months (2nd follow-up)
Illness perception measured with Illness Perception Questionnaire (IPQ) | 9 months (2nd follow-up)
Physical symptoms measured with somatisation subscales from Symptom Check List, 90 items (SCL 90) | 9 months (2nd follow-up)
Health care use (National Patient Register & National Health Service Register (general practitioner (GP) contacts/consultations, specialists, physiotherapists, dentists, GPs' emergency service), The Danish Medicine Agency (medicine consumption)). | 9 months (2nd follow-up)
Sick days (the DREAM database - the register-based evaluation of the extent of marginalization) | 9 months (2nd follow-up)
ACT process measures measured with Five Facet Mindfulness Questionnaire (FFMQ) | 9 months (2nd follow-up)
ACT process measures measured with Acceptance and Action Questionnaire - II (AAQ II) | 9 months (2nd follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Per Fink, DMSc, Study Director — The Research Clinic for Functional Disorders and Psychosomatics, Aarhus University Hospital
Locations (1):
- The Research Clinic for Functional Disorders, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Hoffmann D, Rask CU, Hedman-Lagerlof E, Eilenberg T, Frostholm L. Accuracy of self-referral in health anxiety: comparison of patients self-referring to internet-delivered treatment versus patients clinician-referred to face-to-face treatment. BJPsych Open. 2019 Sep 9;5(5):e80. doi: 10.1192/bjo.2019.54. PMID 31496462
- [Derived] Eilenberg T, Fink P, Jensen JS, Rief W, Frostholm L. Acceptance and commitment group therapy (ACT-G) for health anxiety: a randomized controlled trial. Psychol Med. 2016 Jan;46(1):103-15. doi: 10.1017/S0033291715001579. Epub 2015 Aug 18. PMID 26281857
- See also: Related Info — http://www.functionaldisorders.dk